CLINICAL TRIAL: NCT05284786
Title: Ultrasonographic and Electrophysiological Follow up of Patients With Guillain Barre Syndrome Before and After Treatment
Brief Title: Ultrasonography and Electrophysiology in GBS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Mohammed Galal, specialist, Assiut University
Other Study IDs: ultrasonography in GBS
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Guillain-Barre Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: nerve ultrasonography — Ultrasonography of different nerves was performed using a high frequency 18 MHz probe (esaote Ultrasound systems). Each nerve was scanned in axial plane, and the cross-sectional area (CSA) was measured at standardized anatomical points, in brief: median nerve in upper arm, elbow, forearm; ulnar nerve in upper arm and forearm; tibial nerve in popliteal and ankle; peroneal nerve in popliteal fossa, sural nerve in the calf and the vagus nerve.

SUMMARY:
Description of the time course of nerve ultrasonography changes in correlation to nerve conduction studies (NCS) and clinical course.

DETAILED DESCRIPTION:
GBS is an acute- or subacute-onset polyradiculoneuropathy that often follows an upper or lower respiratory illness or gastroenteritis by 10 to 14 days. Approximately 70% of patients can identify a preceding illness, although it is often benign and may be minimized or forgotten by the patient.

GBS evolves over days, often beginning with numbness in the lower limbs and weakness in the same distribution. The progression of symptoms, particularly weakness, can be rapid, resulting in quadriplegia within a few days. About 50% of patients develop some degree of facial weakness. Weakness attributed to other cranial nerves includes ocular dysmotility, pupillary changes, and ptosis. Thirty percent of patients with GBS develop respiratory failure from phrenic nerve disease, requiring intubation and ventilation. Autonomic involvement is common in GBS, with the most common manifestations being tachycardia, bradycardia, hypertension and hypotension, gastric hypomotility, and urinary retention.

Evidence-based research supports the use of immunotherapy for GBS; proven therapies are IV immunoglobulin (IVIg) and plasma exchange, which have been shown to be equally efficacious in the management of GBS.

At present, no biomarkers exist in the blood, urine, or CSF that confirm the diagnosis of GBS. Most patients with GBS will have an elevated CSF protein, but this laboratory finding may not be present until 3 weeks after the onset of the illness. Nerve conduction studies (NCS) play an important role in support GBS diagnosis and subtype classification. In the first few days of the illness, nerve conduction studies may be normal or only show subtle changes of demyelination, such as prolonged or absent F waves and H reflexes, and patchy changes in distal latencies in patients with AIDP.

More recently, there has been a rise in the use of peripheral nerve ultrasound (US) in the investigation of peripheral neuropathies. Whilst nerve conduction studies (NCS) are helpful at providing information on the function of nerves, US is able to provide information on nerve morphology. The value of nerve ultrasonography (NUS) in immune-mediated polyneuropathies is well described in the previous studies. In post-GBS patients patchy and slight enlargements have been reported. Whereas in acute stage cervical spinal nerve enlargement and hypertrophy of the vagus are probably the most obvious findings. However, only little is known about the course of nerve morphology from onset until clinical recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients newly diagnosed as Guillain Barre Syndrome using diagnostic criteria for GBS.
2. Patients from both sex and at any age group with recent onset of GBS.

Exclusion Criteria:

* Patients with other possible causes of peripheral neuropathy, diabetes, renal, metabolic and others

Ages: 15 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Each patient will be submitted to:
  Clinical assessment scales, ultrasonography assessment of peripheral nerves together with nerve conduction study will performed in all patient within first two weeks of symptoms onset, after two weeks of IVIG or plasmapheresis treatment and after 3 months as follow up.
  1. Comprehensive evaluation at admission with medical history and clinical examination by neurologist.
  2. Clinical assessment scales of different variants GBS:
     1. The overall disability sum score (ODSS).
     2. The Guillain-Barré syndrome disability scale (GDS).
  3. Ultra sonographic assessment of peripheral nerves:
  4. Nerve conduction studies: NCS were performed in the corresponding nerves using a standard electro-neurophysiologic device.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
significance of ultrasonography nerve assessement in follow up of course of the disease | Baseline
  Uses of ultrasonography as an investigatory tool for assessment of changes occur in the nerves over course of disease. Changes in nerves detected by ultrasonography might be an early marker in GBS and support diagnosis of disease in early phase. Also, there are some characteristic differences in ultra-sonographic nerve changes between GBS and CIDP and as known about 15-20% of cases of CIDP are presented with acute onset similar to GBS making an ultrasound can be used as prognostic tool in identification of cases with acute onset CIDP that presented with similar picture of GBS

REFERENCES:
- [Background] Esposito S, Longo MR. Guillain-Barre syndrome. Autoimmun Rev. 2017 Jan;16(1):96-101. doi: 10.1016/j.autrev.2016.09.022. Epub 2016 Sep 23. PMID 27666816
- [Background] van den Berg B, Walgaard C, Drenthen J, Fokke C, Jacobs BC, van Doorn PA. Guillain-Barre syndrome: pathogenesis, diagnosis, treatment and prognosis. Nat Rev Neurol. 2014 Aug;10(8):469-82. doi: 10.1038/nrneurol.2014.121. Epub 2014 Jul 15. PMID 25023340
- [Background] Willison HJ, Jacobs BC, van Doorn PA. Guillain-Barre syndrome. Lancet. 2016 Aug 13;388(10045):717-27. doi: 10.1016/S0140-6736(16)00339-1. Epub 2016 Mar 2. PMID 26948435
- [Background] Asbury AK, Cornblath DR. Assessment of current diagnostic criteria for Guillain-Barre syndrome. Ann Neurol. 1990;27 Suppl:S21-4. doi: 10.1002/ana.410270707. PMID 2194422
- [Background] Hadden RD, Cornblath DR, Hughes RA, Zielasek J, Hartung HP, Toyka KV, Swan AV. Electrophysiological classification of Guillain-Barre syndrome: clinical associations and outcome. Plasma Exchange/Sandoglobulin Guillain-Barre Syndrome Trial Group. Ann Neurol. 1998 Nov;44(5):780-8. doi: 10.1002/ana.410440512. PMID 9818934
- [Background] Uncini A, Kuwabara S. The electrodiagnosis of Guillain-Barre syndrome subtypes: Where do we stand? Clin Neurophysiol. 2018 Dec;129(12):2586-2593. doi: 10.1016/j.clinph.2018.09.025. Epub 2018 Oct 28. PMID 30419502
- [Background] Rajabally YA, Hiew FL, Winer JB. Influence of timing on electrodiagnosis of Guillain-Barre syndrome in the first six weeks: a retrospective study. J Neurol Sci. 2015 Oct 15;357(1-2):143-5. doi: 10.1016/j.jns.2015.07.018. Epub 2015 Jul 14. PMID 26194045
- [Background] Gallardo E, Noto Y, Simon NG. Ultrasound in the diagnosis of peripheral neuropathy: structure meets function in the neuromuscular clinic. J Neurol Neurosurg Psychiatry. 2015 Oct;86(10):1066-74. doi: 10.1136/jnnp-2014-309599. Epub 2015 Feb 4. PMID 25653385
- [Background] Gallardo E, Sedano MJ, Orizaola P, Sanchez-Juan P, Gonzalez-Suarez A, Garcia A, Teran-Villagra N, Ruiz-Soto M, Alvaro RL, Berciano MT, Lafarga M, Berciano J. Spinal nerve involvement in early Guillain-Barre syndrome: a clinico-electrophysiological, ultrasonographic and pathological study. Clin Neurophysiol. 2015 Apr;126(4):810-9. doi: 10.1016/j.clinph.2014.06.051. Epub 2014 Aug 21. PMID 25213352
- [Background] Kerasnoudis A, Pitarokoili K, Behrendt V, Gold R, Yoon MS. Correlation of nerve ultrasound, electrophysiological, and clinical findings in post Guillain-Barre syndrome. J Peripher Nerv Syst. 2013 Sep;18(3):232-40. doi: 10.1111/jns5.12037. PMID 24028191
- [Background] Kerasnoudis A, Pitarokoili K, Behrendt V, Gold R, Yoon MS. Nerve ultrasound score in distinguishing chronic from acute inflammatory demyelinating polyneuropathy. Clin Neurophysiol. 2014 Mar;125(3):635-41. doi: 10.1016/j.clinph.2013.08.014. Epub 2013 Sep 23. PMID 24070674
- [Background] Scheidl E, Bohm J, Simo M, Bereznai B, Bereczki D, Aranyi Z. Different patterns of nerve enlargement in polyneuropathy subtypes as detected by ultrasonography. Ultrasound Med Biol. 2014 Jun;40(6):1138-45. doi: 10.1016/j.ultrasmedbio.2013.12.020. Epub 2014 Mar 5. PMID 24613217
- [Background] Zaidman CM, Al-Lozi M, Pestronk A. Peripheral nerve size in normals and patients with polyneuropathy: an ultrasound study. Muscle Nerve. 2009 Dec;40(6):960-6. doi: 10.1002/mus.21431. PMID 19697380
- [Background] Grimm A, Decard BF, Axer H. Ultrasonography of the peripheral nervous system in the early stage of Guillain-Barre syndrome. J Peripher Nerv Syst. 2014 Sep;19(3):234-41. doi: 10.1111/jns.12091. PMID 25418824